CLINICAL TRIAL: NCT04345588
Title: Comparison of Analgesic Efficacy of Dexamethasone as an Adjuvant in Supraclavicular Block With Intravenous Dexamethasone After Supraclavicular Block in Patients Undergoing Forearm Surgeries
Brief Title: Dexamethasone as an Adjuvant in Supraclavicular Block
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Islam Mohamed Abdel Hamid Ali, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Dexamethasone as an Adjuvant
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Dexamethasone Efficacy as an Adjuvant in Supraclavicular Block
MeSH Terms: interventions — Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: A convenience sample of 60 male and female adult patients will be taken, the patients will be classified into two equal groups , In all patients, we use injection lignocaine 10 mL, injection bupivacaine 0.5% 20 mL, 5 mL normal saline (NS). In one group , injection dexamethasone 0.05 mg/kg will be added to the solution along with IV NS 1cc while the other group will receive 0.05 mg/kg injection dexamethasone intravenously. Duration of analgesia, onset of sensory block, and onset of motor block will be studied.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group received dexamethasone perineural (Active Comparator): injection dexamethasone 0.05 mg/kg perineural.
  Interventions: Drug: Dexamethasone injection
- group received dexamethasone intravenous (Active Comparator): injection dexamethasone 0.05 mg/kg intravenously.
  Interventions: Drug: Dexamethasone injection

INTERVENTIONS:
Drug: Dexamethasone injection — we use injection lignocaine 10 mL, injection bupivacaine 0.5% 20 mL, 5 mL normal saline (NS). In group , injection dexamethasone 0.05 mg/kg will be added to the solution along with IV NS 1cc while the other group will receive 0.05 mg/kg injection dexamethasone intravenously.

SUMMARY:
The use of dexamethasone perineurally along with local anesthetic has been shown to improve the duration of analgesia .

DETAILED DESCRIPTION:
Acute postoperative pain can be effectively controlled with the use of peripheral nerve blocks. Use of additives further prolongs the duration of analgesia For upper limb surgeries below shoulder joint, the brachial plexus block using supraclavicular approach introduced by Kulenkampff has gained popularity. Supraclavicular approach to brachial plexus block is useful for procedures done at or below the level of elbow.

This technique involves the deposition of local anesthetic near the brachial plexus approached from immediately above the clavicle. Brachial plexus is formed by ventral rami of C5, C6, C7, C8, and T1 which forms the roots.These then continue distally to form trunks, divisions, cords,and branches Local anesthetics used alone in supraclavicular block provide analgesia for 4-8 h.

The use of dexamethasone perineurally along with local anesthetic has been shown to improve the duration of analgesia. Intravenous dexamethasone is also useful in attenuating the postoperative need for analgesics in different clinical settings even in the absence of any nerve blocks.

Hence, it is logical to compare the duration of analgesia with the use of dexamethasone in the setting of supraclavicular brachial plexus block, dexamethasone given either perineurally or intravenously.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients between 18 and 60 years of age 2. Both male and female gender 3. ASA physical status Classes I and II patients 4. Patients posted for upper limb surgery below shoulder.

Exclusion Criteria:

* 1. Patient refusal 2. Patients with bleeding disorders and those on anticoagulant therapy 3. History of allergy to local anesthetics 4. Infection at the site of block 5. Neuro deficit involving brachial plexus 6. Pregnant women 7. Patients with psychiatric behavior 8. ASA physical status Classes III and IV patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Dexamethasone efficacy as an Adjuvant in Supraclavicular Block | 2 years
  we will assess the efficacy of dexamethasone in supraclavicular anaethesia in terms of duration of analgesia and onset of motor and sensory block.

CONTACTS AND LOCATIONS:
Overall Officials: Islam Mohamed Abdel Hamid, post graduated, Principal Investigator; Golinar Mohamed Fathy, professor, Study Director; Ahmed Mohamed Abdel Moteleb, lecturer, Study Director

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brummett CM, Williams BA. Additives to local anesthetics for peripheral nerve blockade. Int Anesthesiol Clin. 2011 Fall;49(4):104-16. doi: 10.1097/AIA.0b013e31820e4a49. PMID 21956081
- [Background] Neal JM, Gerancher JC, Hebl JR, Ilfeld BM, McCartney CJ, Franco CD, Hogan QH. Upper extremity regional anesthesia: essentials of our current understanding, 2008. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):134-70. doi: 10.1097/AAP.0b013e31819624eb. PMID 19282714
- [Background] Lalla RK, Anant S, Nanda HS. Verapamil as an Adjunct to Local Anaesthetic for Brachial Plexus Blocks. Med J Armed Forces India. 2010 Jan;66(1):22-4. doi: 10.1016/S0377-1237(10)80086-3. Epub 2011 Jul 21. PMID 27365698
- [Background] Clerc S, Vuilleumier H, Frascarolo P, Spahn DR, Gardaz JP. Is the effect of inguinal field block with 0.5% bupivacaine on postoperative pain after hernia repair enhanced by addition of ketorolac or S(+) ketamine? Clin J Pain. 2005 Jan-Feb;21(1):101-5. doi: 10.1097/00002508-200501000-00012. PMID 15599137
- [Background] Jarbo K, Batra YK, Panda NB. Brachial plexus block with midazolam and bupivacaine improves analgesia. Can J Anaesth. 2005 Oct;52(8):822-6. doi: 10.1007/BF03021776. PMID 16189333
- [Background] Hargreaves KM, Costello A. Glucocorticoids suppress levels of immunoreactive bradykinin in inflamed tissue as evaluated by microdialysis probes. Clin Pharmacol Ther. 1990 Aug;48(2):168-78. doi: 10.1038/clpt.1990.132. PMID 2379387
- [Background] Hong JY, Han SW, Kim WO, Kim EJ, Kil HK. Effect of dexamethasone in combination with caudal analgesia on postoperative pain control in day-case paediatric orchiopexy. Br J Anaesth. 2010 Oct;105(4):506-10. doi: 10.1093/bja/aeq187. Epub 2010 Jul 20. PMID 20659915
- [Background] Movafegh A, Razazian M, Hajimaohamadi F, Meysamie A. Dexamethasone added to lidocaine prolongs axillary brachial plexus blockade. Anesth Analg. 2006 Jan;102(1):263-7. doi: 10.1213/01.ane.0000189055.06729.0a. PMID 16368840
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397
- See also: Iohom G, Machmachi A, Diarra DP, Khatouf M, Boileau S, Dap F, et al.The effects of clonidine added to mepivacaine for paronychia surgery under axillary brachial plexus block. Anesth Analg 2005;100:1179-83. — https://europepmc.org/article/med/15781541
- See also: Comparative Study of Effectiveness of Tramadol and Butorphanol as Adjuvants to Levobupivacaine for Supraclavicular Brachial Plexus Block. — https://europepmc.org/article/PMC/6775833
- See also: Kulenkampff D. Anesthesia of the brachial plexus. Zentralbl Chir 1911;38:1337-40. — https://www.ijss-sn.com/uploads/2/0/1/5/20153321/ijss_mar_oa07_-_2018.pdf